CLINICAL TRIAL: NCT02830659
Title: Cochlear Implants Registry in Thailand Project
Acronym: CIRT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Khon Kaen University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Kwanchanok Yimtae, M.D., Director of Neuro-otology unit, Khon Kaen University
Other Study IDs: HE591146; HSRI. 59-031 (Other Grant/Funding Number: Health System Research Institution); CERT004/59BRm (Other: Central Research Ethics Committee)
Record Dates: First submitted 2016-07-02; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Cochlear Implantation

STUDY DESIGN:
Observational Model: Case-Only

SUMMARY:
The purpose of this study is to determine the outcome of cochlear implant including post operative hearing ability, developing of language, complication from cochlear implant, quality of life, and success factor of cochlear implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery with cochlear implant

Exclusion Criteria:

* Patients who reject to participate with this project

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who underwent surgery for cochlear implant
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Aids Threshold 1 | 1 year
  The pure tone air-conduction threshold at 0.25, 0.5, 1, 2, 3, 4, 6, 8 kilohertz, measuring in the sound-proof room using the standard audiometry while patient is using cochlear implants.

SECONDARY OUTCOMES:
CAP 1 | 1 year
  Categories of Auditory Performance (CAP) is an index consisting of eight performance categories, relating to auditory perception. It is arranged in a hierarchy of skills that increase in difficulty for example from the ability to perceive environmental sounds right up to using the telephone. It is widely used in the range of current research on children with cochlear implants and is an easy to use tool for monitoring progress.
Quality of life | 5 years
  The quality of life will be assessed by interviewing questionnaires using HUI-3.

CONTACTS AND LOCATIONS:
Locations (11):
- Thailand (11):
  - King Bhumibol Adulyadej Hospital, Bangkok, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok, Bangkok
  - Department of Otolaryngology Phramongkutklao College of Medicine, Bangkok, Bangkok
  - Rajavithi Hospital, Bangkok, Bangkok
  - Ramathibodi Hospital, Bangkok, Bangkok
  - Siriraj Hospital, Bangkok, Bangkok
  - Department of Otolaryngology, Srinakharinwirot University, Bangkok, Bangkok
  - Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen
  - Songkhlanagarind Hospital, Songkhla, Changwat Songkhla
  - Trang Hospital, Trang, Changwat Trang
  - Department of Otolaryngology, Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai